CLINICAL TRIAL: NCT00255671
Title: Prospective Study on the Short-Term Adverse Effects From Gamma Knife Radiosurgery
Brief Title: Acute Side Effects in Patients Who Are Undergoing Stereotactic Radiosurgery for Brain Tumors or Other Brain Disorders
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE4Z05
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer; Radiation Toxicity
Keywords: radiation toxicity; tumors metastatic to brain; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic meningioma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult diffuse astrocytoma; adult ependymoblastoma; adult ependymoma; adult giant cell glioblastoma; adult gliosarcoma; adult medulloblastoma; adult melanocytic lesion; adult meningeal hemangiopericytoma; adult meningioma; adult myxopapillary ependymoma; adult oligodendroglioma; adult papillary meningioma; adult pineoblastoma; adult pineocytoma; adult subependymoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult mixed glioma; recurrent adult brain tumor; adult pilocytic astrocytoma; adult glioblastoma; ACTH-producing pituitary tumor; growth hormone-producing pituitary tumor; nonfunctioning pituitary tumor; prolactin-producing pituitary tumor; recurrent pituitary tumor; TSH producing pituitary tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Radiation Injuries; Brain Neoplasms; Astrocytoma; Ependymoma; Meningioma; Oligodendroglioma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Medulloblastoma; Pinealoma; Glioma, Subependymal; Glioma; Growth Hormone-Secreting Pituitary Adenoma; Pituitary Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Determine the incidence and types of acute complications in patients undergoing stereotactic radiosurgery for brain tumors or other brain disorders.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Questionnaire — Patients complete questionnaires about the side effects they experience from radiosurgery. The questionnaires are completed at baseline and at 1 week, 1 month, and 2 months after radiosurgery.

SUMMARY:
RATIONALE: Learning about the side effects of stereotactic radiosurgery in patients with brain tumors or other brain disorders may help doctors plan treatment and help patients live more comfortably.

PURPOSE: This clinical trial is studying the acute side effects in patients who are undergoing stereotactic radiosurgery for brain tumors or other brain disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence and types of acute complications in patients undergoing stereotactic radiosurgery for brain tumors or other brain disorders.
* Determine the time frame for development and resolution of these complications in these patients.
* Determine the severity of these complications in these patients.

OUTLINE: Patients undergo stereotactic radiosurgery. Patients also complete questionnaires about the side effects they experience from radiosurgery. The questionnaires are completed at baseline and at 1 week, 1 month, and 2 months after radiosurgery.

PROJECTED ACCRUAL: A total of 94 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of brain tumor or other brain disorder, including, but not limited to, 1 of the following:

  * Primary brain tumors
  * Brain metastases
  * Acoustic neuromas
  * Pituitary adenomas
  * Parkinson's disease
  * Cluster headaches
  * Glomus jugulare
  * Epilepsy
  * Obsessive compulsive disorder
  * Arteriovenous malformations
  * Trigeminal neuralgia
* Eligible for and scheduled to undergo stereotactic radiosurgery

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No physical or mental limitation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Endocrine therapy

* Concurrent steroids allowed

Radiotherapy

* No prior stereotactic radiosurgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Short-term adverse effects as assessed by a questionnaire | at 1 week, 1 month, and 2 months
  Patients undergo stereotactic radiosurgery. Patients also complete questionnaires about the side effects they experience from radiosurgery. The questionnaires are completed at baseline and at 1 week, 1 month, and 2 months after radiosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: John Suh, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States